CLINICAL TRIAL: NCT03969199
Title: Give a MANNA a Fish, Teach a MANNA to Fish
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 829424
Record Dates: First submitted 2019-05-22; First posted 2019-05-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Cirrhosis, Liver; Liver Diseases; Malnutrition
Keywords: MANNA; Nutrition; Cirrhosis, Liver; Liver Diseases; Dietary compliance; Low sodium diet; Non-profit; Salt affinity; Behavioral changes
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Malnutrition | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MANNA Food Delivery Service (Experimental): MANNA will deliver meals to patients randomized to the intervention arm of the study every week on the same day for 90 days. Each delivery will include: 7 breakfast meals, 7 lunch meals, 7 dinner entrees, health desserts, and fresh fruit. Meals will be delivered frozen and can be stored in a freezer until ready to eat. Patients will be followed for 180 days and will be assessed for their salt affinity and urine sodium at 3 separate time points throughout the study: baseline, 90 days, and 180 days.
  Interventions: Behavioral: Intervention
- Standard of Care Counseling (No Intervention): Patients randomized to the control arm will receive standard or care dietary counseling from either their physician or a dietician. Patients will be followed for 180 days and will be assessed for their salt affinity and urine sodium at 3 separate time points throughout the study: baseline, 90 days, and 180 days.

INTERVENTIONS:
Behavioral: Intervention — Dietary intervention in coordination with MANNA, who will deliver low sodium meals to patients for 90 days
  Arms: MANNA Food Delivery Service

SUMMARY:
This study is a randomized pilot seeking to address low patient adherence to a low sodium diet as a strategy to improve outcomes of patients with cirrhosis of the liver. In coordination with the Metropolitan Area Neighborhood Nutrition Alliance (MANNA) of Philadelphia, patients in the intervention cohort will receive low sodium MANNA meals to encourage improved dietary compliance. Outcomes of these interventional patients will be compared to those receiving standard of care--namely, educational intervention by physicians supplemented by occasional counseling from dieticians during clinic visits encouraging a low sodium diet. Dietary compliance will be evaluated by urine sodium and salt affinity tests and used as a positive marker for improved outcomes. The target population of this study is patients diagnosed with cirrhosis of the liver, aged 18-85 years living within the MANNA-serviced area.

DETAILED DESCRIPTION:
Malnutrition causes and complicates numerous chronic illnesses. One in three hospitalized patients in the United States is malnourished, accounting for delayed recovery, increased complications, extended length of stay, and avoidable utilization of healthcare. The projected cost of chronic disease from 2016-2030 in Pennsylvania is $1.7 trillion, with 5% of people accounting for 50 % of healthcare spending.

Patients with cirrhosis of the liver often present with profound malnutrition due to the catabolic effects of their disease. Because of this, adhering to a low sodium diet is of paramount importance in order to avoid fluid overload, a common cause for hospital readmission of patients with cirrhotic decompensations. By maintaining a proper diet, it is possible to mitigate the medical deterioration of patients as well as mitigate the expense of managing chronic illnesses like cirrhosis.

Results from MANNA, a not-for-profit food delivery service, have shown a monthly care cost reduction for patients receiving meals from $41,000 to $28,000, and monthly inpatient cost reduction from $220,000 to $132,000. Results also show that changes in nutritional behavior also improve treatment rates, physical activity, and reduce substance abuse. MANNA has been able to deliver more than 13,000,000 meals to over 20,000 clients since 1990. 99% of patients reported improved overall health after receiving the meals, 92% reported improved emotional health, 98% said it reduced their stress, and 96% said the meals improved their energy. Existing solutions in most health systems are nutritional counseling (either very briefly by a physician, or if patients are fortunate, by a dietician). This is usually not a longitudinal process, and patients are often overwhelmed by medical information.

Despite their remarkable results the acute illness space (6 months of meals), the MANNA service is not scalable to the management of chronic illness; through this study investigators seek to bridge that gap. In coordination with MANNA, investigators will provide 3 months of low sodium MANNA meals to patients in the interventional cohort in an effort to encourage improved adherence to a low sodium diet. Dietary compliance will be assessed using urine sodium and salt affinity tests, and results will be compared between the cohort receiving MANNA meals and the cohort receiving standard of care dietary counseling. Investigators will continue to follow patients for an additional 3 months following the completion of their MANNA service to determine if receiving pre-made low sodium meals for even a short period of time is likely to provide any long-term benefit beyond the span of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cirrhosis of the liver
* 18 to 85 years old
* Ability to read and provide informed consent
* Resides in an area serviced by MANNA
* Has a medical need for restriction of dietary sodium

Exclusion Criteria:

* Unclear diagnosis of cirrhosis of the liver
* Inability to provide informed consent
* Any other reason for which the investigator feels the participant would be unable to safely follow the study protocol.
* Resides in an area not serviced by MANNA
* Nutritional needs that cannot be accommodated by MANNA (i.e. vegan or vegetarian, nut-free, gluten-free, Kosher, Macrobiotics and/or allergy to milk, eggs, soybean, peanuts, tree nuts, fish and shellfish.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Differential adherence to a low sodium diet during intervention | 90 days
  A measurable difference in dietary compliance during participation in the MANNA meal program. Compliance will be assessed by performing urine sodium analyses coupled with salt affinity tests following the first 90 days of the study.

SECONDARY OUTCOMES:
Sustained differential adherence to low sodium diet following intervention | 180 days
  A measurable maintained difference in dietary compliance after MANNA meal delivery ceases. Compliance will be assessed by performing urine sodium analyses coupled with salt affinity tests following the final 90 days of the study after MANNA delivery has ended for the intervention arm.